CLINICAL TRIAL: NCT03761407
Title: A Phase-I Study to Investigate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Multiple Escalating Oral Doses of GRT0151Y in Healthy Male and Female Subjects
Brief Title: A Clinical Study in Healthy Subjects Which Aims to Investigate the Safety, the Tolerability and the Effects of GRT0151Y and How the Compound is Taken up and Excreted From the Body
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Grünenthal GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HP0151Y/09
Record Dates: First submitted 2018-11-30; First posted 2018-12-03 (Actual); Last update posted 2018-12-03 (Actual); Status verified 2018-11

CONDITIONS: Acute Pain
MeSH Terms: conditions — Acute Pain

STUDY DESIGN:
Intervention Model Description: Twelve volunteers (6 males and 6 females) per dose group will be randomly assigned to two treatment sequences (placebo-verum and verum-placebo, within dose-group randomized) in a ratio of 1:1. There will be a washout period of 7 to 11 days between the treatment sequences.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1 (100 mg GRT0151Y) (Experimental): The dose of 100 mg will be administered twice (b.i.d.) on Day 1 (titration day). On Days 2, 3 and 4, the treatment regimen will be changed to a triple daily (t.i.d) medication with 100 mg. On Day 5 the last dose of 100 mg will be administered in the morning.
  Matching placebo using the same dosing regimen as defined in the treatment group.
  Interventions: Drug: 100 mg GRT0151Y; Drug: Matching placebo
- Group 2 (125 mg GRT0151Y) (Experimental): The dose of 125 mg will be administered twice (b.i.d.) on Day 1 (titration day). On Days 2, 3 and 4, the treatment regimen will be changed to a triple daily (t.i.d) medication with 125 mg. On Day 5 the last dose of 125 mg will be administered in the morning.
  Matching placebo using the same dosing regimen as defined in the treatment group
  Interventions: Drug: 125 mg GRT0151Y; Drug: Matching placebo
- Group 3 (150 mg GRT0151Y) (Experimental): The dose of 150 mg will be administered twice (b.i.d.) on Day 1 (titration day). On Days 2, 3 and 4, the treatment regimen will be changed to a triple daily (t.i.d) medication with 150 mg. On Day 5 the last dose of 150 mg will be administered in the morning.
  Matching placebo using the same dosing regimen as defined in the treatment group
  Interventions: Drug: 150 mg GRT0151Y; Drug: Matching placebo
- Group 4 (225 mg GRT0151Y) (Experimental): The dose of 150 mg will be administered twice (b.i.d.) on Day 1 (titration day). On Days 2, 3 and 4, the dose of 225 mg will be administered twice (b.i.d.). On Day 5 the last dose of 225 mg will be administered in the morning.
  Matching placebo using the same dosing regimen as defined in the treatment group
  Interventions: Drug: 225 mg GRT0151Y; Drug: Matching placebo

INTERVENTIONS:
Drug: 100 mg GRT0151Y — 100 mg capsule (1 x 100 mg capsule)
  Arms: Group 1 (100 mg GRT0151Y)
Drug: 125 mg GRT0151Y — 125 mg (1 x 100 mg capsule and 1 x 25 mg capsule)
  Arms: Group 2 (125 mg GRT0151Y)
Drug: 150 mg GRT0151Y — 150 mg (1 x 100 mg capsule and 1 x 50 mg capsule)
  Arms: Group 3 (150 mg GRT0151Y)
Drug: 225 mg GRT0151Y — Day 1: 150 mg (1 x 100 mg capsule and 1 x 50 mg capsule) Day 2 - 5: 225 mg (2 x 100 mg capsules and 1 x 25 mg capsule)
  Arms: Group 4 (225 mg GRT0151Y)
Drug: Matching placebo — Matching placebo capsules using the same dosing regimen as defined in the treatment groups.

SUMMARY:
The aim of this clinical study in healthy participants is to investigate the safety and tolerability of GRT0151Y after multiple oral intake of different increasing doses and to evaluate the pharmacological effects (action of the compound) by means of pupillometry (measuring the pupil size of the eye) and Cold Presser Test (measuring the pain when immersing the hand in 2 degree Celsius cold water). An additional aim of the study is to investigate the pharmacokinetics of GRT0151Y (how it is taken up into the body and how it is excreted from the body)."

ELIGIBILITY:
Inclusion Criteria:

* Male or female Caucasian.
* Age 40-65 years.
* Body mass index (BMI) between 18 and 30 kilograms/square meter (extremes included).
* Extensive Cytochrome P450 2D6 (CYP2D6) metabolizer.
* Healthy as determined by medical history, physical examination, vital signs, 12-lead electrocardiogram (ECG), and clinical laboratory parameters (haematology, Blood sedimentation rate (BSR), clotting, bio-chemistry, urinalysis and virus serology). Minor deviations of laboratory values and ECG parameters from the normal range may be accepted, if judged by the investigator as clinically not relevant and if not considered to interfere with the study objectives.
* Adequate contraception. For females of childbearing potential (i.e. all females except surgically sterilized or at least 2 years postmenopausal) this is defined as follows: any form of hormonal contraception or intra-uterine device must be used, at least for 4 weeks prior to the first dosing AND she must give a consent to use an additional barrier contraception (condom or diaphragm) from 2 weeks prior to first dosing up to 4 weeks after the last dosing.
* Written consent to participate in the study.
* Negative Human immunodeficiency virus (HIV)1/2-antibodies, Hepatitis B surface (HBs)-antigen, Hepatitis B core (HBc)-antibodies, Hepatitis C virus (HCV)-antibodies determined at screening examination.
* Negative drug abuse screening test determined at screening examination (the test will include screening for metamphetamine, opiate, cannabis, cocaine, amphetamine and benzodiazepine).
* Negative beta-human chorion gonadotropin test for females of childbearing potential determined at screening examination (the test is not necessary in females who are in post-menopausal state for at least 2 years or in females with status after surgical sterilisation).
* The participant must be able to tolerate the cold pressor test, i.e. he/she must be able to keep his/her hand for 120 seconds in cold water of about 2 degrees celsius.
* The participant must be able to undergo the procedure of pupillometry.

Exclusion Criteria:

* Pulse rate below 45 or above 100 Beats per minute (bpm). The measurement must be performed in supine position after a resting period of at least 5 minutes.
* Systolic blood pressure below 100 or above 160 Millimeter mercury (mmHg), diastolic blood pressure below 50 or above 100 mmHg. The measurement must be performed in supine position after a resting period of at least 5 minutes.
* History or presence of diseases or functional disorders of the Central nervous system (CNS), endocrinological system, gastrointestinal tract, hepatobiliary system, renal system, respiratory system or cardiovascular system or other conditions known to interfere with the absorption, distribution, metabolism or excretion of drugs.
* Marked repolarisation abnormality (e.g. suspicious or definite congenital long QT syndrome) or co-medication that is known to influence cardiac repolarisation substantially.
* History of seizures or at risk (epilepsy in family anamnesis, unclear loss of consciousness), head trauma requiring hospitalization.
* Neurotic personality, psychiatric illness or suicide risk.
* History of orthostatic hypotension.
* Bronchial asthma.
* Definite or suspected history of drug allergy or hypersensitivity.
* History of Raynaud´s disease or phenomenon.
* Malignancy.
* Participation in another clinical study within three month prior to the start of this study (exception: characterization of metabolizer status).
* Blood donation (more than 100 Milliliter(s) or a comparable blood loss within three month prior to the start of this study.
* Excessive consumption of food or beverages containing caffeine or other xanthines (more than 1000 Milliliter(s) coffee or equivalent per day) within two weeks prior to the start of this study.
* Evidence of alcohol, medication or drug abuse.
* Smokers who are not able to abstain from smoking during the hospitalisation.
* Intake of drugs that are inhibitors of CYP2D6 isoenzyme within the last 4 weeks prior to the start of this study. Use of any other medication within two weeks prior to the start of the study (self-medication or prescription), if not on a stable basis and known to interfere with study objectives.
* Known or suspected of not being able to comply with the study protocol or of not being able to communicate meaningfully with the investigator and staff.
* Opinion of the investigator the volunteer should not participate in the study.
* Pregnant or breastfeeding.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2004-12-30 (Actual); Primary Completion 2005-07-26 (Actual); Study Completion 2005-07-26 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events. | From the first IMP administration (Day 1) to the Final Examination (Day 4 to 11 after last period).
  Number of adverse events and number of participants with adverse events.

SECONDARY OUTCOMES:
Pupillometry parameter: Initial pupil diameter | Day 1 at 0 hour, 4, 11 and 23 hours, on Day 2 at 11 and 23 hours and on Day 5 at 0 hour, 1 hour, 4, 11, 23, 35 and 47 hours
  Pupil size (in mm) will be measured using a Compact Integrated Pupillograph (CIP). Measurements will be performed always in the same eye of the individual (preferably the left eye). The measurements will be performed under standard low-light conditions (10-15 lux).
Pupillometry parameter: Amplitude of constriction | Day 1 at 0 hour, 4, 11 and 23 hours, on Day 2 at 11 and 23 hours and on Day 5 at 0 hour, 1 hour, 4, 11, 23, 35 and 47 hours
  Amplitude of constriction (difference between initial pupil diameter and minimum pupil diameter [mm])
Pupillometry parameter: Onset latency of miosis | Day 1 at 0 hour, 4, 11 and 23 hours, on Day 2 at 11 and 23 hours and on Day 5 at 0 hour, 1 hour, 4, 11, 23, 35 and 47 hours
  Onset latency of miosis (the time between begin of light stimulus and the onset of constriction [ms])
Pupillometry parameter: Constriction time | Day 1 at 0 hour, 4, 11 and 23 hours, on Day 2 at 11 and 23 hours and on Day 5 at 0 hour, 1 hour, 4, 11, 23, 35 and 47 hours
  Constriction time (time for maximum pupil contraction [s])
Minimum plasma concentration during dosing interval τ at steady-state (Css,min) | predose on Day 1, during 4 consecutive days of multiple dosing and up to 72 hours after the last dosing on Day 5
Maximum plasma concentration during dosing interval τ at steady-state (Css,max) | predose on Day 1, during 4 consecutive days of multiple dosing and up to 72 hours after the last dosing on Day 5
Time to reach maximum plasma concentration during dosing interval τ at steady-state (tss,max) | predose on Day 1, during 4 consecutive days of multiple dosing and up to 72 hours after the last dosing on Day 5
Area under the concentration vs. time curve after the last dose (AUC) | predose on Day 1, during 4 consecutive days of multiple dosing and up to 72 hours after the last dosing on Day 5
Average plasma concentration during dosing interval τ at steady-state (Css,ave) | predose on Day 1, during 4 consecutive days of multiple dosing and up to 72 hours after the last dosing on Day 5
Peak-trough fluctuation at steady-state (PTF%) | predose on Day 1, during 4 consecutive days of multiple dosing and up to 72 hours after the last dosing on Day 5
Rate constant for the terminal log-linear phase of the concentration time data, computed as the negative slope of the regression line for the terminal linear phase of the logarithmic concentration versus time plot (λss,z) | predose on Day 1, during 4 consecutive days of multiple dosing and up to 72 hours after the last dosing on Day 5
Half-life for the terminal log-linear phase of the concentration time data (tss,1/2,z) | predose on Day 1, during 4 consecutive days of multiple dosing and up to 72 hours after the last dosing on Day 5
Apparent terminal half-life after last dose (t1/2,Z) | predose on Day 1, during 4 consecutive days of multiple dosing and up to 72 hours after the last dosing on Day 5
Apparent terminal elimination rate constant after last dose (λz) | predose on Day 1, during 4 consecutive days of multiple dosing and up to 72 hours after the last dosing on Day 5
Area under the concentration vs. time curve in dosing interval τ at steady-state (AUCss,τ) | predose on Day 1, during 4 consecutive days of multiple dosing and up to 72 hours after the last dosing on Day 5
Extrapolated part to infinity of AUCss at steady-state (AUCextr) | predose on Day 1, during 4 consecutive days of multiple dosing and up to 72 hours after the last dosing on Day 5
Extrapolated part to infinity of AUCss in percent at steady-state (AUC%extr) | predose on Day 1, during 4 consecutive days of multiple dosing and up to 72 hours after the last dosing on Day 5
Area under the concentration-time data for dosing interval τ (AUC0-τ) | predose on Day 1, during 4 consecutive days of multiple dosing and up to 72 hours after the last dosing on Day 5
Total mean time in the total volume of distribution (MRTvsys) | predose on Day 1, during 4 consecutive days of multiple dosing and up to 72 hours after the last dosing on Day 5
Relative total clearance (CL/F)ss | predose on Day 1, during 4 consecutive days of multiple dosing and up to 72 hours after the last dosing on Day 5
Relative volume of distribution for the terminal log-linear phase of the concentration time data (Vz/F)ss | predose on Day 1, during 4 consecutive days of multiple dosing and up to 72 hours after the last dosing on Day 5
Cold Pressor Test (CPT) (AUC of pain assessment) | Day 1 at 0 hour, 4, 11 and 23 hours, on Day 2 at 11 and 23 hours and on Day 5 at 0 hour, 1, 4, 11, 23, 35 and 47 hours.
  The dominant hand will be plunged into a 1-3 degrees Celsius circulating cold water quench for 2 minutes. By using a computer mouse with the other hand, the participant adjusted a visual analogue scale on a computer screen facing them. The scale was labelled "no pain" at one end and "maximum pain" at the other end.

CONTACTS AND LOCATIONS:
Overall Officials: Grünenthal Study Director, Study Director — Grünenthal GmbH
Locations (1):
- ASTER, Paris, France

IPD SHARING:
Plan to Share IPD: No